CLINICAL TRIAL: NCT00912990
Title: Pediatric Elective Intubation With and Without Muscle Relaxation Utilizing the Shikani Optical Stylet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adequate subjects numbers not enrolled in study timeframe.
Sponsor: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Sandeep Khanna, Attending Physician Division of Pediatric Critical Care, Rady Children's Hospital, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11672; 06104C (Other: Rady Children's Hospital San Diego)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Intubation,Endotracheal
Keywords: Pediatric
MeSH Terms: interventions — cisatracurium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Placebo Comparator): Normal saline volume calculated to be equal to the volume of cisatracurium 0.2mg/kg
  Interventions: Drug: Normal saline
- Cisatracurium (Active Comparator): Subjects in this arm will be given Cisatracurium 0.2mg/kg IV dose one time prior to intubation.
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — One intravenous dose: 0.2mg/kg/dose
  Other Names: Nimbex
  Arms: Cisatracurium
Drug: Normal saline — One Intravenous dose
  Arms: Normal saline

SUMMARY:
The investigators' primary specific aims are to demonstrate that:

1. Pediatric patients with normal airways, undergoing elective surgical procedures, can be successfully intubated when deeply sedated, without the use of muscle relaxants using the Shikani Optical Stylet.
2. Shikani intubation of pediatric patients is equally effective in children that are deeply sedated or paralyzed as evidenced by a non-significant difference in:

   * Time to intubation (defined as no more than a 30 second time difference between the two groups);
   * Incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 6 months of age to 17 years of age (not yet 18)
* Male or female
* English or Spanish speaking
* Normal airway (Mallampati Classification )
* American Society of Anesthesiology Physical Status Classification I or II
* Elective surgical procedure expected to last at least 45 minutes in length
* Written informed consent/assent for participation given by the parent legal guardian and subject (if applicable)

Exclusion Criteria:

* < 6 months of age, > 17 years of age
* Difficult airway (Mallampati Classification)
* History of previous difficult intubation, suspected abnormal airway: *micrognathia

  * facial trauma
  * airway tumor
  * epiglottitis
  * retropharyngeal abscess
  * foreign body, etc.
  * Scheduled for non-elective, emergent OR procedure
  * Parent, legal guardian, or subject is unavailable or unwilling to consent for study participation

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at a single, pediatric hospital site.
Groups:
- Cisatracurium: Subjects in this arm will be given Cisatracurium 0.2mg/kg IV dose one time prior to intubation.
  Cisatracurium : One intravenous dose: 0.2mg/kg/dose
- Normal Saline: Normal saline volume calculated to be equal to the volume of cisatracurium 0.2mg/kg
  Normal saline : One Intravenous dose
Period: Overall Study
Arm/Group | Cisatracurium | Normal Saline
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisatracurium | Normal Saline | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: Time to intubation was defined as the time (seconds) required to verify three breaths on an end-tidal carbon dioxide monitor.
Time Frame: Confirmed by the visualization of three carbon dioxide waveforms.
Population: Unable to summarize data or complete analysis due to small study sample and technical problems with measurement leading to unreliable data.
Arm/Group | Cisatracurium | Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Number of Adverse Events
Description: The number of occurrences of each event. One subject may have multiple adverse events.
Time Frame: Recorded from the start of the intubation procedure to the time of successful endotracheal intubation
Population: No further statistical analysis (intent-to-treat) completed due to small study sample.
Measure: Number; unit: events
Arm/Group | Cisatracurium | Normal Saline
Number analyzed (Participants) | 16 | 18
events | 0 | 3

3. Other Pre Specified Outcome: Number of Intubation Attempts for Each Enrolled Subject
Description: The total number of intubation attempts to achieve successful intubation of study participants.
Time Frame: The number is totaled after successful endotracheal intubation is documented
Population: Unable to analyze data due to small study sample.
Arm/Group | Cisatracurium | Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cisatracurium | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisatracurium (N=16) | Normal Saline (N=18)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Participant movement/cough/gag (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Inadequate subject numbers led to early termination. Unable to adequately power the study for data analysis. OAE data reported for transparency only and should not be used to extrapolate significant conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No